CLINICAL TRIAL: NCT05950438
Title: A Prospective Clinical Registry Investigating Outcomes of Elective Robotic Transhiatal Esophagectomy
Brief Title: Investigating Outcomes of Elective Robotic Transhiatal Esophagectomy
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ankit Bharat, Chief of Thoracic Surgery, Northwestern University
Other Study IDs: STU00219267
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Esophagectomy
Keywords: Robotic Transhiatal
MeSH Terms: interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy is a complex surgical procedure performed to treat various esophageal disorders. The surgery involves the removal of all or part of the esophagus and reconstruction using other parts of the gastrointestinal tract.

SUMMARY:
The primary goal of this study is to collect short-term and long-term health outcomes of a robotic transhiatal esophagectomy procedure. Clinical (or health) outcomes measure the effect of the procedure on your overall health status. During this procedure, the surgeon will remove all or part of your esophagus. We want to identify patients who will have this procedure. We will look at data elements before, during, and after your procedure to understand the impact of this surgery on your post-operative clinical outcomes.

DETAILED DESCRIPTION:
Esophagectomy is a complex surgical procedure performed to treat various esophageal disorders. The surgery involves the removal of all or part of the esophagus and reconstruction using other parts of the gastrointestinal tract. Different surgical approaches and techniques have been developed, including open (transthoracic or transhiatal), minimally invasive (video-assisted thoracoscopic surgery or robotic-assisted), and hybrid approaches. These techniques may yield different clinical outcomes, and there is still ongoing debate regarding the optimal approach. Nevertheless, minimally invasive approaches, including robotic esophagectomy, are generally preferred given the lower morbidity. This prospective clinical registry aims to investigate outcomes of elective robotic transhiatal esophagectomy, the preferred approach at Northwestern Memorial Hospital, for adult patients undergoing this procedure. By collecting clinical and demographic data prospectively, we hope to identify factors that contribute to improved outcomes and guide future surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Patients undergoing elective esophagectomy for any indication
* Patients who have already had an elective esophagectomy for any indication
* Patients with consent providing capacity

Exclusion Criteria:

* Patients undergoing emergent esophagectomy
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Vulnerable Populations

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified in the Thoracic Surgery clinic or in the inpatient setting based on the surgeon's expertise who need to undergo an elective esophagectomy procedure.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Anastomotic Leak | During first 3 months postop
  Postoperative Complication
Number of Participants with Esophageal Stricture | During first 3 months postop
  Postoperative Complication
Number of Participants with Pneumonia | During first 3 months postop
  Postoperative Complication
Number of Participants Requiring Ventilation >48 Hours | During first 3 months postop
  Postoperative Complication
Number of Participants with Empyema | During first 3 months postop
  Postoperative Complication
Number of Participants with Pulmonary Embolism | During first 3 months postop
  Postoperative Complication
Number of Participants with Deep Venous Thrombosis | During first 3 months postop
  Postoperative Complication
Number of Participants with Gastric Outlet Obstruction | During first 3 months postop
  Postoperative Complication
Number of Participants with Stroke | During first 3 months postop
  Postoperative Complication
Number of Participants with Atrial Fibrillation | During first 3 months postop
  Postoperative Complication
Number of Participants with Vocal Cord Paralysis | During first 3 months postop
  Postoperative Complication
Number of Participants with Myocardial Infarction | During first 3 months postop
  Postoperative Complication
Number of Participants with Chylothorax | During first 3 months postop
  Postoperative Complication
Number of Participants with Acute Renal Injury | During first 3 months postop
  Postoperative Complication
Number of Participants with Wound Infections | During first 3 months postop
  Postoperative Complication
Rates of Re-operation | During first 3 months postop
  Postoperative Complication
Rates of Re-Admission | During first 3 months postop
  Postoperative Complication
Number of Participants with Intensive Care Unit (ICU) Stay | During first 3 months postop
  Postoperative Complication
Rates of Length of Hospital Stay | Postoperative
  Postoperative Complication
Rates of 30-day Survival | Postoperative
  Postoperative Complication
Rates of 90-day Survival Rates | Postoperative
  Postoperative Complication

SECONDARY OUTCOMES:
Operative Time of Surgery | Intraoperative
  Length of Surgery
Rates of Blood Loss | Intraoperative
  Did the Participant Lose Any Blood During the Surgery
Number of Participants with Conversion Rates to Open Esophagectomy | Intraoperative
Number of Participants with Lymph nodes in the Final Specimen | Intraoperative
  Pathological Variables
Number of Participants with Proximal and Distal Margins | Intraoperative
  Pathological Variables

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Bharat, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No